CLINICAL TRIAL: NCT04942184
Title: Improving Memory in Daily Life of Patients With Alzheimer's Disease
Brief Title: STRATEGIES to Improve Memory in Alzheimer's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started due to the Covid 19 pandemic.
Sponsor: Boston University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-40597; P30AG013846 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer Disease; Dementia, Mild; Mild Cognitive Impairment
Keywords: Memory; Memory Strategies; EEG headgear
MeSH Terms: conditions — Alzheimer Disease; Dementia; Lymphoma, Follicular; Cognitive Dysfunction | interventions — Electroencephalography; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1- 15 Mild AD and 15 MCI due to AD (Experimental): In Group 1, for the first 2 weeks participants will be taught memory strategies and reminded to use them each day from week 0 to week 2. Weeks 3-4, participants will be advised to keep using the strategies both on the tablet and in their daily life even though they will not be reminded each time they start the task.
  Interventions: Behavioral: Memory strategies in Arm 1; Device: Electroencephalogram (EEG) headset in Arm 1; Other: Tablet in Arm 1
- Group 2- 15 Mild AD and 15 MCI due to AD (Active Comparator): In Group 2, for the first 2 weeks participants will be reminded to "try hard" to remember the items although they will not be given any specific strategies. At week 2 the subjects will be taught memory strategies and reminded to use them each day from week 2 to week 4.
  Interventions: Behavioral: Memory strategies in Arm 2; Device: Electroencephalogram (EEG) headset in Arm 2; Other: Tablet in Arm 2

INTERVENTIONS:
Behavioral: Memory strategies in Arm 1 — Memory strategies will consist of daily at-home exercises lasting between 20 minutes to 1 hour depending on the memory tasks assigned to each participant. At the start of week 1 participants will be taught the memory strategies to use while completing the daily memory tasks. In week 1 and 2, subjects will be reminded daily to use the memory strategies. At the start of week 3, subjects will be advised to use the memory strategies however they will not be given daily reminders.
  Arms: Group 1- 15 Mild AD and 15 MCI due to AD
Device: Electroencephalogram (EEG) headset in Arm 1 — A cap that measures brain activity using a 16-sensor wireless dry (no gel applied) EEG device designed by BrainWaveBank Ltd., that uses Bluetooth technology to securely transmit EEG signals to an Android tablet. The cap will be used during week 1,2,3 and 4.
  Arms: Group 1- 15 Mild AD and 15 MCI due to AD
Other: Tablet in Arm 1 — A computer tablet will be provided to each participant that will have daily reminders about the memory strategies during week 1 and 2, while no reminders will be present in week 3 and 4. The tablet software includes a user-friendly interface that provides feedback and instructions that help the participant properly wear the EEG headset. At the end of each session the tablet stores behavioral and EEG data on a secured server accessible by the research staff.
  Arms: Group 1- 15 Mild AD and 15 MCI due to AD
Behavioral: Memory strategies in Arm 2 — Memory strategies will consist of daily at home exercises lasting between 20 minutes to 1 hour depending on the memory tasks assigned to each participant. During weeks 1 and 2, participants will be completing the memory tasks without being instructed to use any specific strategy. At the end of week 2 subjects will be taught the memory strategies and during week 3 and 4, they will be reminded daily to use the memory strategies while completing the memory tasks.
  Arms: Group 2- 15 Mild AD and 15 MCI due to AD
Device: Electroencephalogram (EEG) headset in Arm 2 — A cap that measures brain activity using a 16-sensor wireless dry (no gel applied) EEG device designed by BrainWaveBank Ltd., that uses Bluetooth technology to securely transmit EEG signals to an Android tablet. The cap will be used during week 1,2,3 and 4.
  Arms: Group 2- 15 Mild AD and 15 MCI due to AD
Other: Tablet in Arm 2 — A computer tablet will be provided to each participant. During week 3 and 4, the tablet will present daily reminders to use memory strategies while completing the memory tasks. The tablet software includes a user-friendly interface that provides feedback and instructions that help the participant properly wear the EEG headset. At the end of each session the tablet stores behavioral and EEG data on a secured server accessible by the research staff.
  Arms: Group 2- 15 Mild AD and 15 MCI due to AD

SUMMARY:
Memory mistakes are one of the most detrimental symptoms in Alzheimer's Disease (AD). In this study the investigators will measure the long-term efficacy of memory strategies in patients with AD. First, the efficacy of the strategies will be evaluated in the laboratory by analyzing the behavioral response and the brain activity of the patients. During the first visit, patients will be taught the memory strategies and asked to repeat them at home for 4 weeks. During this period of time, patients will perform several memory tasks while their performance and brain activity will be measured using portable devices. Monitoring brain activity and behavioral responses to memory tasks will provide insightful information on the efficacy of the strategies and allow the investigation of how patients can maintain the strategies over time. The research will examine if improving memory through the use of cognitive strategies, can positively affect other domains of daily life.

DETAILED DESCRIPTION:
A crossover design with two groups will be implemented to test the following objectives:

Primary Objective: To determine the long-term efficacy of memory strategies in AD patients using experimental memory paradigms and standard neuropsychological tests. Over the course of 4 weeks, performance on novel memory tasks and standard neuropsychological tests will evaluate the efficacy of the strategies longitudinally.

Secondary Objectives:

1. To determine the neural mechanism of memory strategies in AD patients through portable electroencephalogram/event-related potential (EEG/ERP) electrophysiology. Portable EEG will allow us to measure the electrophysiological changes associated with the use of memory strategies over time during daily life of patients with AD.
2. To determine how memory strategies, influence the daily life and functioning of the AD patients. Questionnaires on daily life activities will be administered at different timepoints to determine whether patients are able to generalize the strategies to tasks in their daily life.

This research study will investigate whether the use of combined memory strategies (conservative and deep/item-specific encoding) can help improve performance in memory tasks, can be maintained over time, and can be generalized to other tasks in daily life. Depending on the study group, either at week 0 visit or week 2 visit, participants will be trained on the two strategies. A power point presentation will be used to display one example of each of the strategies and how to implement them during the tablet/Ipad tasks. At this time the investigators will answer any other specific questions that might come up about the strategies. Before starting the cognitive tasks at home on the app, the tablet will remind participants about using the strategies, and this will also include an example how the strategies should be implemented.

The two memory strategies will be implemented in the described steps below:

While being presented with a list of items (words or objects), participants will be asked to focus on one unique characteristic of the items (item-specific encoding strategy). Afterwards, another list of items, containing previously studied (old) and unstudied (new) items, will be presented. Participants will be asked to recognize whether the item was presented in the previous list and respond "yes" only if they are absolutely sure of their response (conservative strategy). Participants will then be provided with a number of real-world examples to practice generalizing what they have learned.

ELIGIBILITY:
Inclusion Criteria:

For Mild Alzheimer Disease (AD) dementia

* meets probable AD dementia National Institute on Aging and Alzheimer's Association (NIA-AA) criteria
* Mini-Mental State Examination (MMSE) 20-27
* performance on delayed recall and recognition memory worse than 1.5 standard deviation (SD) for age and education
* performance on delayed recall and recognition memory worse than 1.5 SD for age & education in at least one other cognitive domain (e.g., language, executive functioning) based on other tests in our neuropsychological test battery.
* Dr. Turk and Dr. Budson will confirm all mild AD dementia diagnoses

For Mild cognitive impairment (MCI)

* meets MCI due to AD NIA-AA criteria
* MMSE > 23
* performance on delayed recall and recognition memory worse than 1.0 SD for age & education adjusted norms
* Dr. Turk and Dr. Budson will confirm all MCI due to AD diagnoses

Exclusion Criteria:

A clinically significant problem of any of the following conditions:

* depression
* heavy alcohol or drug use
* cerebrovascular disease
* traumatic brain damage
* a different degenerative disease (e.g., fronto-temporal dementia, Parkinson's disease)
* any medical condition whose severity could significantly impair cognition (e.g., organ failure)
* Unable to understand the consent form

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in performance in memory tasks over time | baseline, 4 weeks
  Change in performance in memory tasks will be measured through daily at home memory exercises that will last from 20 minutes to 1 hour. Higher the scores on the exercise represent better memory performance.

SECONDARY OUTCOMES:
Change in electroencephalogram (EEG) early negative frontal component (N400) | Baseline, 4 weeks
  Change in EEG early negative frontal component (N400) will be assessed by measuring amplitude and latency characteristics of this EEG component. A higher amplitude and shorter latency will show improvement in memory performance.
Change in EEG Late Positive Parietal Component (LPC) | Baseline, 4 weeks
  Change in EEG Late Positive Parietal Component (LPC) will be assessed by measuring amplitude and latency characteristics of this EEG component. A higher amplitude and shorter latency will show improvement in memory performance.
Change in EEG Late Positive Frontal Effect (LFE) | Baseline, 4 weeks
  Change in EEG Late Positive Frontal Effect (LFE) will be assessed by measuring the amplitude and latency characteristics of this EEG component. A higher amplitude and shorter latency will show improvement in memory performance.
Neuropsychological assessment using the Montreal Cognitive Assessment (MoCA) | baseline, 4 weeks
  Neuropsychological assessment will be completed using the Montreal Cognitive Assessment (MoCA).
  The MoCA has a total score of 30, and a higher score means improved cognitive performance.
Neuropsychological assessment using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). | Baseline, 4 weeks
  Neuropsychological assessment will be completed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). The RBANS has a total index score of 160, and it measures performance in the following domains: immediate memory, visuospatial, language, attention, and delayed memory. A higher score on the RBANS means improved cognitive performance.
Generalization of strategies to daily life functioning | Baseline, 4 weeks
  Generalization of strategies will be assessed through the Activities of Daily Living Scale (ADL) which is a 31-item questionnaire assessing the ability to complete activities of daily living. The minimum score is 0 while the maximum score is 279. A lower score on the Activities of Daily life scale means a greater level of independence in completing activities of daily life.
Quality of life with Alzheimer's disease | Baseline, 4 weeks
  Quality of life will be assessed with the Quality of Life in Alzheimer's Disease (QoLAD) which is a 13-item questionnaire assessing different aspects of quality of life. The minimum score is 13 and the maximum is 52. A higher score represents better quality of life.
Subjective perception of memory performance | Baseline, 4 weeks
  Subjective perception of memory performance will be assessed using the Multifactorial Metamemory Questionnaire (MMQ), which is a 61-item questionnaire divided in three subcategories (Contentment, Ability and Strategy). The minimum score is 0 and the maximum is 244. A higher score means a better subjective memory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Turk, MD, Principal Investigator — BU School of Medicine

IPD SHARING:
Plan to Share IPD: No